CLINICAL TRIAL: NCT01632800
Title: Sensory Effects of Rapidly-Changing Magnetic Fields
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weinberg Medical Physics LLC (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: WMP 5.0; R42HL086294-04 (NIH); 9R42NS073289-06 (NIH)
Record Dates: First submitted 2010-03-17; First posted 2012-07-03 (Estimated); Results first posted 2016-06-15 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Sensory Disorders
Keywords: Magnetic fields discomfort
MeSH Terms: conditions — Sensation Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm study (Experimental): Each subjects will undergo escalating exposure to magnetic field
  Interventions: Device: High pulsed magnetic fields

INTERVENTIONS:
Device: High pulsed magnetic fields — Magnetic fields will escalate in strength
  Other Names: Pulser is custom built by Applied Pulsed Power, Ithaca NY

SUMMARY:
This study is being conducted to improve magnetic resonance imaging (MRI) scans by reducing the time required for imaging. Experience has shown that unpleasant side-effects from magnetic pulses used in MRI (for example, tingling or tapping sensations) can be reduced when the magnetic pulses are shortened. In this study, we will explore whether this effect holds true when very short magnetic pulses are applied.

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18, capable of informed consent

Exclusion Criteria:

* History of arrhythmia. Has implanted pacemaker or defibrillator, right wrist-to-sternum distance of less than 60 centimeters, visible tattoos of the right hand or wrist, or with any metallic objects that cannot be removed from the right hand or wrist. Irregular or imperceptible pulse. Heart rate less than 50 beats per minute or more than 100 per minute, resting respiratory rate greater than 25 per minute, diastolic blood pressure less than 50. Solid meal ingested within 2 hours prior to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Fricke, PhD, Principal Investigator — Children's National Research Institute
Locations (1):
- Applied Pulsed Power, Freeville, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm Study
Started | 26
Completed | 25
Not Completed | 1
Not completed — Subject did not fit in apparatus | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Study
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Degree of Discomfort Under Applied Pulsed Magnetic Fields
Description: Pulsed magnetic fields will be applied a total of forty-eight times to the right hand of each subject. After each time the magnet coil is pulsed, the subject will be asked if he or she notices any sensation (for example, tingling or tapping). Subjects will be asked to rate the sensation from 0 to 4, where 0 means no sensation, 1 means barely-noticeable sensation, 2 means easily noticeable sensation, 3 means unpleasant sensation, and 4 means very unpleasant sensation.
Time Frame: Bioeffects will be assessed within the five-minute application of each pulse sequence
Measure: Number; unit: percentage of subjects with discomfort
Arm/Group | Single Arm Study
Number analyzed (Participants) | 25
percentage of subjects with discomfort | 0

ADVERSE EVENTS:
Arm/Group | Single Arm Study
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes